CLINICAL TRIAL: NCT01647464
Title: Study of Whether There is Renal Retention of Lipid Microbubble Ultrasound Contrast Agents
Brief Title: Renal Retention of Microbubbles
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor of Medicine, Oregon Health and Science University
Other Study IDs: MBretention
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: - Study Focus: Renal Retention of Lipid Microbubbles

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Contrast administration: Patients undergoing contrast-enhanced echo.

SUMMARY:
Flank pain has been reported with ultrasound (US) contrast agents. The purpose of this study is to determine whether there is retention of ultrasound contrast agents in the renal microcirculation, which has been described in mice.

DETAILED DESCRIPTION:
In this study patients undergoing clinically indicated contrast echocardiography will have renal ultrasound performed 10 minutes after completion of contrast infusion to determine the presence and location of renal retention of lipid microbubbles.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing clinically indicated contrast echo
* adequate renal ultrasound images

Exclusion Criteria:

* chronic inflammatory disease
* known kidney disease
* immunomodulatory therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing contrast echocardoigraphy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrast Administration
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects undergoing contrast echo
Arm/Group | Contrast Administration
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Renal Video Intensity Units
Description: Video intensity units in the kidney 10 min after completion of a clinically indicated contrast echocardiography study.
Time Frame: 10 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contrast Administration
Number analyzed (Participants) | 10
units on a scale | 19 (9)

ADVERSE EVENTS:
Arm/Group | Contrast Administration
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No